CLINICAL TRIAL: NCT05484869
Title: Comparison of Perinatal and Neonatal Outcomes of Very Advanced Maternal Aged Pregnants and Early Adolescent Pregnant Women
Brief Title: Very Advanced Maternal Aged Pregnants and Early Adolescent Pregnant Women
Status: Completed | Type: Observational
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Serif Aksin, associate professor, Siirt University
Other Study IDs: SiirtUNIVER
Record Dates: First submitted 2022-07-22; First posted 2022-08-02 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Advanced Maternal Age Pregnancy; Early Pregnancy
Keywords: age; pregnancy; adolescent; perinatal; neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early Adolescent Pregnant Women (n:80): Perinatal and neonatal results of adolescent pregnancies of 16 years and below
- Very Advanced Maternal Aged Pregnants (n:67): Perinatal and neonatal results of pregnancies 45 years and older
- Reproductive period Control Group (n:150): Reproductive period Pregnant Between 25-35 years

SUMMARY:
Maternal age is an important factor affecting the pregnancy process and its results. Adverse obstetric outcomes such as preterm birth, stillbirth, and infant mortality are more common in women older than 35 years and younger than 20 years compared to women aged 20-29. Adolescent pregnancies have been associated with an increased risk of adverse pregnancy outcomes such as preterm birth, low birth weight, perinatal death, and maternal mortality.

Advanced maternal age pregnancies were associated with higher rates of maternal hypertension and diabetes, and progressively worsening perinatal outcomes such as stillbirth, preterm birth, and low birth weight.

Although the investigators' region has high birth rates, as far as they have observed, the rates of early and advanced maternal age are also quite high. the investigators' aim in this study is to determine the absolute effects of early and advanced maternal age on pregnancy and to investigate the pregnancy outcomes of these mothers.

DETAILED DESCRIPTION:
The investigators' aim in this study is to determine the absolute effects of early and advanced maternal age on pregnancy and to investigate the pregnancy outcomes of these mothers. For this purpose, the information of 90 pregnant women followed in Siirt Training and Research Hospital between 2017-2021 will be accessed through the hospital's data system. Maternal age, pregnancy history, Assisted reproductive technologies history, laboratory findings, screening test results, mode of delivery, baby birth information, pregnancy complications and complications during delivery will be recorded. In the light of the information gathered, the rates of negative effects of gestational age on pregnancy will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnants under the age of 16 and younger
* pregnants over the age of 45 and older

Exclusion Criteria:

* history of chronic hypertension
* history of pre gestational diabetes
* history of chronic diseases
* excessive consumption of alcohol
* smoking pregnants
* kidney disorders

Ages: 15 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant on the age of 16 and below and on the age of 45 and above, control groups
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Delivery type in pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  The % of delivery type (vaginal delivery/ cesarean section) will be compared between the three groups
Abortion ratio of pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of abortion will be compared between the three groups
Neonatal death ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of neonatal death will be compared between the three groups
Premature rupture of membranes in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of premature rupture of membranes (PROM) will be compared between the three groups
Preterm labor ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of preterm labor will be compared between the three groups
Ablatio placentae ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of ablatio placentae will be compared between the three groups
Fetal Distress ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of fetal distress will be compared between the three groups
Intrauterine death ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of intrauterine death will be compared between the three groups
Gestational diabetes ratio in pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of gestational diabetes mellitus (GDM) will be compared between the three groups
Preeclampsia ratio in pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of preeclampsia will be compared between the three groups
Surmaturation ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of surmaturation will be compared between the three groups
Polyhydramnios ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of polyhydramnios will be compared between the three groups
Oligohydramnios ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of oligohydramnios will be compared between the three groups
Presentation anomaly ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of presentation anomaly will be compared between the three groups
Multiple pregnancy ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of multiple pregnancy will be compared between the three groups
Intrauterine growth retardation ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of intrauterine growth retardation (IUGR) will be compared between the three groups
Postpartum hemorrhage ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of postpartum hemorrhage will be compared between the three groups
Placenta previa ratio in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  Rate and % of placenta previa will be compared between the three groups
Mean fetal weight of pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1month
  The fetal weight (in grams) will be compared between the three groups
Ratio of male, female gender in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  % of male, female gender will be compared between the three groups
Mean APGAR scores in the 1st minute in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  APGAR scores in the 1st minute (by numbers) will be compared between the three groups
Mean APGAR scores in the 5th minute in pregnancies of pregnant women under the age of 16 ( group 1), over the age of 45 (group 2) and between the age of 25-35 (group 3). | 1 month
  APGAR scores in the 5th minute (by numbers) will be compared between the three groups

CONTACTS AND LOCATIONS:
Overall Officials: Şerif Aksin, Assoc.Prof, Study Director — Siirt University Medical Faculty Obstetrics and Gynecology Departmant

REFERENCES:
- [Background] Brown W, Ahmed S, Roche N, Sonneveldt E, Darmstadt GL. Impact of family planning programs in reducing high-risk births due to younger and older maternal age, short birth intervals, and high parity. Semin Perinatol. 2015 Aug;39(5):338-44. doi: 10.1053/j.semperi.2015.06.006. Epub 2015 Jul 10. PMID 26169538
- [Background] Malabarey OT, Balayla J, Klam SL, Shrim A, Abenhaim HA. Pregnancies in young adolescent mothers: a population-based study on 37 million births. J Pediatr Adolesc Gynecol. 2012 Apr;25(2):98-102. doi: 10.1016/j.jpag.2011.09.004. Epub 2011 Nov 16. PMID 22088316
- [Background] Traisrisilp K, Tongsong T. Pregnancy outcomes of mothers with very advanced maternal age (40 years or more). J Med Assoc Thai. 2015 Feb;98(2):117-22. PMID 25842790